CLINICAL TRIAL: NCT02261792
Title: Parallel Randomised Open Blind Evaluation Study of the Efficacy of 20° Trendelenburg Position During 24 Hours After Epidural Blood Patch in the Treatment of Spontaneous Intracranial Hypotension
Brief Title: Spontaneous Intracranial Hypotension Treatment "SIHT"
Acronym: SIHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P111118; 2013-AO1017-38 (Other: IDRCB)
Record Dates: First submitted 2014-09-26; First posted 2014-10-10 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Spontaneous Intracranial Hypotension
Keywords: Postural headache treatment; Spontaneous intracranial hypotension; Epidural blood patch; Trendelenburg position; Head-Down Tilt; Blood Patch, Epidural
MeSH Terms: conditions — Intracranial Hypotension | interventions — Head-Down Tilt; Bed Rest; Blood Patch, Epidural

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A : 24 hours bed rest (Active Comparator): 24 hours bed rest
  Interventions: Procedure: 24 hours bed rest; Procedure: EBP
- B : 24 hours Trendelenburg position (Experimental): 24 hours Trendelenburg position
  Interventions: Procedure: 24 hours Trendelenburg position; Procedure: EBP

INTERVENTIONS:
Procedure: 24 hours Trendelenburg position — Trendelenburg position
  Other Names: inclination of the body at 20 degrees
  Arms: B : 24 hours Trendelenburg position
Procedure: 24 hours bed rest — 24 hours bed rest after EBP
  Other Names: Allitement flat position for 24 hours
  Arms: A : 24 hours bed rest
Procedure: EBP — Autologous Epidural Blood Patch
  Other Names: Epidural Blood Patch

SUMMARY:
Spontaneous intracranial hypotension (SIH) is an infrequent disease, related to a leak of cerebrospinal fluid. There are not controlled studies for this treatment.The main of this study is to demonstrate the superiority of the Trendelenburg position compared to supine position during 24 hours after an epidural blood patch for a spontaneous intracranial hypotension

DETAILED DESCRIPTION:
Various treatments have been used for patient with spontaneous intracranial hypotension, but there is not definite approach. Some patients, fortunately, improve spontaneously. Bed rest and increased fluid intake have been advocate. The effectiveness of the caffeine has been shown in some studies, but durable beneficial effect is doubtful. The efficacy of steroids has not been established. However, although there have been no controlled studies, autologous epidural blood patch (EBP) can be considered the treatment of choice for patients. The success rate of EBP for a post lumbar puncture headache is about 90%, but for SIH, is very less about 50% after the first one and 77% after the second. The amount of blood injected must be sufficient. On the other hand, the leak is usually located on dorsal, above the prolonged rest must be respected. One study, have demonstrated, without randomization, a success rate of 90% with a prolonged Trendelenburg after EBP. We decided to do this study, to confirm a superiority of a 24 hours prolonged Trendelenburg position.

It's a monocentric study of parallel randomized open blind groups. Patients will be recruited by investigators in our headache emergency room. If the diagnose of SIH is confirmed (orthostatic headache from more than 5 days and less than 28 days with a normal MRI or with sign of SIH) study will be proposed.

After a signed information, the patients will be randomized in 2 groups, the investigator is blind of the randomized arm of patient

1. EBP with 24 hours bed rest
2. EBP with 24 hours Trendelenburg position

V1: inclusion V2 : 24 hours before EBP (headache, associated symptoms, HIT6) V3 : randomization and EBP V4 : first evaluation 30 minutes after standing (headaches, associated symptoms) V5 : phone evaluation (safety) D7 V6 : Evaluation at D15 (headache, associated symptoms, safety) V7 : Evaluation at D30 (headache, associated symptoms, control cerebral MRI, HIT6, safety) V8 : last evaluation D60 (headache, associated symptoms,HIT6 safety)

Collection of 2nd EBP, 3rd EBP, 4th EBP throughout the study up to J 92 maximum

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* No contraindication for BPE
* Severe or moderate headache within 15 min standing, mild or no headache after 15 min bed rest
* Headache from 5 to 28 days
* Normal or evidence of low CSF on MRI
* Signed informed consent

Exclusion Criteria:

* Known dural leak in the previous 2 months the onset of headache
* Abnormal MRI
* First BPE for SIH
* The patient has participated in another clinical trial than can interact with the evaluation
* Contraindication of Trendelenburg position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Recovery at Day 1 without relapse at Day 15 | Day 1
  V4: first evaluation 30 minutes after standing (headaches, associated symptoms) V6 : Evaluation at D15 (headache, associated symptoms, safety)
Recovery at Day 1 without relapse at Day 15 | day 15
  V4: first evaluation 30 minutes after standing (headaches, associated symptoms) V6 : Evaluation at D15 (headache, associated symptoms, safety)

SECONDARY OUTCOMES:
2d EBP and other EBP | day 7, 15, 30 and 60
  Number of patients requires a treatment with a second BP at any time of study (withdrawal study)
Associated symptoms | day 1, 15, 30 and 60
  Disappearance of associated symptoms
Headache | day 1,15, 30 and 60
  Pain scores, localisation and type of persistent headache at day 1,15, 30 and 60
subdural hematoma surgery | day 7, 15, 30 and 60
  Number of patients requires a surgery for life-threatening acute SDH
cerebral MRI | day 30
  results of D30 control MRI, compared to baseline MRI
medullar MRI | day 60
  results of baseline medullar MRI and the link between leak and patient recovery
Epidural Blood Patch | day 60
  Volume of blood and localisation of injection / statistical data related with recovery

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROOS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Lariboisiere Hospital - Centre Urgences Céphalées (CUC), Paris, France

REFERENCES:
- [Background] Ferrante E, Arpino I, Citterio A, Wetzl R, Savino A. Epidural blood patch in Trendelenburg position pre-medicated with acetazolamide to treat spontaneous intracranial hypotension. Eur J Neurol. 2010 May;17(5):715-9. doi: 10.1111/j.1468-1331.2009.02913.x. Epub 2009 Dec 29. PMID 20050898
- [Background] Sencakova D, Mokri B, McClelland RL. The efficacy of epidural blood patch in spontaneous CSF leaks. Neurology. 2001 Nov 27;57(10):1921-3. doi: 10.1212/wnl.57.10.1921. PMID 11723293